CLINICAL TRIAL: NCT01049230
Title: Phase II Study of Proton Radiation Therapy for CNS Germ Cell Tumors: Evaluation of Acute and Late Side Effects
Brief Title: Proton Beam Radiation Therapy for Central Nervous System (CNS) Germ Cell Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kevin X. Liu, MD, DPHIL, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-263
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Germ Cell Tumor; Central Nervous System Germ Cell Tumor
Keywords: proton beam radiation; CNS germ cell tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton beam radiation (Experimental): Radiation therapy with proton beam
  Interventions: Radiation: Proton Beam radiation

INTERVENTIONS:
Radiation: Proton Beam radiation — Once a day, 5 days a week (Monday-Friday), for 4-8 weeks

SUMMARY:
The purpose of this research study is to determine if radiation using proton beam therapy will kill the germ cell tumor in the participant's central nervous system. This type of radiation has been used previously on many patients with different types of cancers. There are two types of external radiation treatments, proton beam and photon beam. In this study we will be examining the effects of proton beam radiation therapy. Studies have suggested that this kind of radiation can spare normal tissue more than photon radiation therapy. The physical characteristics of proton beam radiation let the doctor safely increase the amount of radiation delivered to the tumor. We believe that proton beam therapy will potentially reduce side effects that participants would normally experience with photon radiation therapy.

DETAILED DESCRIPTION:
* Before participants begin radiation therapy they will have scans done to prepare them for radiation treatment. Doctors will use the information gathered from these scans to plan the best way to deliver radiation to the tumor.
* Participants will receive treatment as an outpatient at the Francis H. Burr Proton Center located at the Massachusetts General Hospital.
* Not everyone who participates in this study will receive the same amount of proton radiation therapy. The length of time and amount of radiation that the participant will receive will depend on the type of germ cell tumor they have and the stage of the their disease.
* Radiation treatment will be given once a day, 5 days a week (Monday-Friday), for 4-8 weeks depending on the condition of the participant's disease.
* During each week of proton radiation therapy, participants will have a physical exam and be asked questions about their general health and any problems they might be experiencing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed germ cell tumor or elevated AFP or B-HCG in the setting of radiographic disease consistent with a germ cell tumor. Disease must be confined to the central nervous system.
* Participants do not need to have measurable disease. Most patients will not have measurable disease at the time of treatment.
* 3 years of age or older and 25 years of age or younger at the time of diagnosis because this study evaluates this disease entity in the pediatric population which may differ from the adult population.
* Life expectancy of greater than 12 months.
* ECOG performance status of 0, 1 or 2
* Baseline MRI of the brain and spinal axis with gadolinium and prior to any chemotherapy is required. If surgical resection is performed a post-operative MRI is required. If the patient receives chemotherapy prior to radiation, a post-chemotherapy MRI of the brain is required. If spinal involvement was seen on initial MRI and prior to chemotherapy, a MRI of the spine is required after chemotherapy and prior to radiation.
* Serum and lumbar CSF must be obtained to evaluate for alpha fetoprotein (AFP) and beta human chorionic gonadotropin (HCG). This is needed to stratify patients into pure GCT and NGGCT.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients will be ineligible if any prior therapeutic radiation therapy > 200 cGy has been delivered to the central nervous system.
* Patients will be ineligible if chemotherapy was completed greater than 1 year from the planned start date of radiation therapy or if the patient is referred for radiation therapy after a relapse following a regimen with chemotherapy alone.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals diagnosed and treated within the past 5 years for cervical cancer in situ and basal cell or squamous cell carcinoma of the skin.
* Pregnant females

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To describe late complications of craniospinal, whole ventricle, and involved field radiation therapy delivered with proton radiotherapy in place of photon radiation for this patient population. | 2 years
To evaluate acute and subacute toxicities of craniospinal, whole ventricle, and involved field radiation therapy delivered with proton radiotherapy in place of photon radiation in this patient population. | 2 years

SECONDARY OUTCOMES:
To determine 3 year progression free survival rate of patients with pure germ cell tumors and non-germinomatous germ cell tumors treated with proton radiation. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shannon MacDonald, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts